CLINICAL TRIAL: NCT00929955
Title: Study of Role of Anti-Inflammatory Agents in Patients With Schizophrenia
Brief Title: Role of Anti-Inflammatory Agents in Patients With Schizophrenia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pakistan Institute of Living and Learning (Other)
Collaborators: Karwan e Hayat (Unknown); Dow University of Health Sciences (Other)
Responsible Party: Dr Imran B Chaudhry, University of Manchester
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PILL-UoM-0110
Record Dates: First submitted 2009-06-28; First posted 2009-06-30 (Estimated); Last update posted 2019-08-05 (Actual); Status verified 2019-08

CONDITIONS: Schizophrenia; Schizoaffective Disorder; Psychosis Not Otherwise Specified; Schizophreniform Disorder
Keywords: Anti inflammatory; Schizophrenia; Simvastatin; ondansetron
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Ondansetron; Simvastatin

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Ondansetron (Active Comparator)
  Interventions: Drug: Ondansetron
- Simvastatin (Active Comparator)
  Interventions: Drug: Simvastatin
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ondansetron — ondansetron added to TAU Ondansetron will be administered in 8mg once daily dose
  Arms: Ondansetron
Drug: Simvastatin — Simvastatin added to TAU Simvastatin 20mg taken as once daily dose
  Arms: Simvastatin
Drug: Placebo — Placebo added to TAU
  Arms: Placebo

SUMMARY:
There is some evidence that anti-inflammatory treatment may have beneficial effects in schizophrenia and major depression. Cox-2 inhibitors have been tested in preliminary clinical trials for schizophrenia and depression, showing favourable effects compared to placebo (Muller and Schwarz et al 2009).

Statins were introduced as cholesterol-lowering agents but have found much wider usage. They are anti-inflammatory agents and thus similar to the Cox-2 inhibitors, which have shown some ability as adjuncts to improve the symptoms of schizophrenia in preliminary studies. The statins are also known to decrease C-reactive protein (CRP), which has been shown in an SMRI-funded study to be elevated in a study of individuals with schizophrenia. Fan et al (2007) demonstrated in a small study in patients with schizophrenia that higher than normal levels of CRP (>0.50 mg/dl) was associated with marked negative symptoms and higher total PANSS scores.

Ondansetron is a serotonin (5-HT3) receptor antagonist that is generic and widely used to prevent nausea and vomiting in patients receiving chemotherapy for cancer. GSK did a small study on it as an antipsychotic in the 1980s. Since then, several small studies have suggested that it is effective as an adjunct drug in improving the symptoms of schizophrenia.

Statins are widely used in schizophrenia sufferers, particularly those taking second generation antipsychotics, to treat hypercholesterolemia. Both drugs are well tolerated and their side effect profiles well understood.

We propose to conduct a feasibility study in patients with chronic schizophrenia to explore the adjunct use of simvastatin and ondansetron on positive, negative and general psychopathology in comparisons to treatment as usual (TAU) over a 12 week period.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnostic and Statistical Manual-IV (DSM-IV) diagnosis of schizophrenia, schizoaffective disorder, psychosis not otherwise specified or schizophreniform disorder
2. competent and willing to give informed consent
3. stable on medication 4 weeks prior to baseline
4. able to take oral medication and likely to complete the required evaluations
5. female participants of child bearing age must be willing to use adequate contraceptives for the duration of the study, and, willing to have a pregnancy test pre treatment and at ten weekly intervals while on study medication.

Exclusion Criteria:

1. Relevant medical illness [renal and hepatic] in the opinion of the investigators
2. history of high alcohol intake
3. any change of psychotropic medications within the previous six weeks
4. diagnosis of substance abuse (except nicotine or caffeine) or dependence within the last three months according to DSM-IV criteria
5. pregnant or breast-feeding.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2009-06 (Actual); Primary Completion 2009-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
acceptability and tolerability of simvastatin and ondansetron added to TAU | 3 months

SECONDARY OUTCOMES:
simvastatin and ondansetron added to TAU prevents the accumulation of negative symptoms in patients with schizophrenia | 3 months
simvastatin and ondansetron added to TAU prevents cognitive decline | 3 months
To compare the effect size | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Imran B Chaudhry, MD, Principal Investigator — University of Manchester
Locations (2):
- Pakistan (2):
  - Dow University of Health Sciences, Karachi
  - Karwan e hayat, Karachi